CLINICAL TRIAL: NCT02955381
Title: 6 Month Double-Blind Randomized Placebo-Controlled Trial to Evaluate the Safety and Efficacy of Small Particle Hyaluronic Acid to Treat Acne Scars Located on the Cheeks and Forehead
Brief Title: Restylane Silk Acne Scar Efficacy Evaluation Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Liquidation of Research Department
Sponsor: Schweiger Dermatology, PLLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SDG 02-2016
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Acne; Acne Scars; AdverseEvent
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Restylane Silk, 1.0 ml (Experimental): Subjects must have at least 1 but up to 3 acne scars ≥3 mm and ≤ 10 mm located on the cheeks or forehead. Subjects will receive one treatment (Restylane® Silk) in each scar (up to 3 acne scars) at day 0, and Month 1 (2 total treatments per scar during the study). Subjects will remain blinded to the treatment administered to them during these visits.
  Interventions: Device: Restylane Silk, 1.0 ml
- Placebo (Saline), 1.0 ml (Placebo Comparator): Subjects must have at least 1 but up to 3 acne scars ≥3 mm and ≤ 10 mm located on the cheeks or forehead. Subjects will receive one treatment (Placebo (Saline)) in each scar (up to 3 acne scars) at day 0, and Month 1 (2 total treatments per scar during the study). Subjects will remain blinded to the treatment administered to them during these visits.
  Interventions: Device: Saline, 1.0 ml

INTERVENTIONS:
Device: Restylane Silk, 1.0 ml — Restylane® Silk was approved in 2014 submucosal implantation for lip augmentation and dermal implantation for correction of perioral rhytids in patients over the age of 21.
  Arms: Restylane Silk, 1.0 ml
Device: Saline, 1.0 ml — Simple saline solution. To be used as placebo (control). No active ingredients.
  Arms: Placebo (Saline), 1.0 ml

SUMMARY:
Randomized, double-blind, placebo-controlled, research pilot study. 30 subjects aged 22-55 years old of all skin types will be asked to sign an informed consent form prior to any study procedures. Subjects must have at least 1 but up to 3 acne scars ≥3 mm or ≤ 10 mm located on the cheeks or forehead. Subjects will receive one treatment (Restylane® Silk or Placebo) in each scar at day 0, and Month 1 (2 total treatments per scar during the study). Subjects will be asked to come to 10 visits: Screening visit (up to 35 days prior to Baseline), Baseline (Day 0), Day 7, Day 14, Month 1, Month 2, Month 3, Month 4, Month 5, and Month 6 (study exit visit). The treatment area will be evaluated at each visit by the unblinded investigator regarding erythema, bruising, inflammation, itching, stinging/burning, brightness, fullness, smoothness, and clarity. Safety and adverse events will be captured at each visit only by the unblinded investigator.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, research pilot study. 30 subjects aged 22-55 years old of all skin types will be asked to sign an informed consent form prior to any study procedures. Subjects must have at least 1 but up to 3 acne scars ≥3 mm or ≤ 10 mm located on the cheeks or forehead. Subjects will receive one treatment (Restylane® Silk or Placebo) in each scar at day 0, and Month 1 (2 total treatments per scar during the study). Subjects will be asked to come to 10 visits: Screening visit (up to 35 days prior to Baseline), Baseline (Day 0), Day 7, Day 14, Month 1, Month 2, Month 3, Month 4, Month 5, and Month 6 (study exit visit). The blinded investigators will evaluate the target scar using the Acne Scar Rating Scale (ASRS), rate the target acne scar regarding treatment effect on a -5 ("Markedly worse"), to 0 ("Neutral Improvement"), to 5 (Markedly Improved (Clear or nearly clear)) point scale, and evaluate the skin quality (regarding brightness, fullness, smoothness, and clarity). Subjects will give the acne scar a score on the subject VAS acne scar satisfaction scale marking between 0 ("Not satisfied with Acne Scar at Day 0") and 10 ("Extremely Satisfied with Acne Scar at Day 0"). The treatment area will be evaluated at each visit by the unblinded investigator regarding erythema, bruising, inflammation, itching, stinging/burning, brightness, fullness, smoothness, and clarity. The subject will have their vital signs taken, complete a symptom diary (only if the subject experiences side effects or adverse events), complete a DLQI, and have photos (VECTRA and 2D digital photographs) taken of the treatment area. Efficacy measures will only be completed by the blinded investigator. Safety and adverse events will be captured at each visit only by the unblinded investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female subjects on an acceptable form of birth control aged 22-55 years of age.
2. Willing to refrain from undergoing any procedures to repair or augment any acne scar in the treatment area during the study.
3. Female subjects with a negative pregnancy test confirmed at screening and on an acceptable form of birth control. Acceptable forms of birth control on this study include oral or injectable contraceptive, contraceptive patches, Depo-Provera, NuvaRing, Implanon, double barrier methods, IUD, same sex partner, or abstinence. Males will be required to use an acceptable method of birth control: vasectomy, double-barrier method, condom with spermicidal lube, or abstinence.
4. Signed informed consent prior to conducting any study procedures.
5. Willing to refrain from undergoing any cosmetic procedures in the treatment area during the study.
6. At least one acne scar located on the cheeks or forehead to be ≥ 3 mm and ≤ 10 mm in diameter, and rated as ≥3 on the ASRS at day 0. Subjects may have up to three qualifying acne scars determined eligible for treatment at screening.
7. Acne scars that are classified as either ice pick, rolling, or boxcar acne scars.
8. ≤15 pustules/papules on the face at the time of screening and ≤ 2 nodules, and no cysts at Baseline.
9. Willing to attend all study visits and comply with protocol

Exclusion Criteria:

1. Subjects with active cystic acne at screening (> 2 nodules or any cysts present at Baseline).
2. Use of antibiotics 2-weeks prior to screening.
3. Use of retinoids 2-weeks prior to screening.
4. Use of salicylic acid or benzoyl peroxide 7 days prior to screening.
5. Excessive facial hair, skin conditions, facial tattoos, or other dermatologic marks that would obscure the treatment area.
6. Use of Isotretinoin (Accutane) 6 months prior to screening.
7. Semi-permanent or permanent injection in the face 3 months prior to screening.
8. History of bleeding disorders.
9. Use of blood thinners (i.e warfarin (Coumadin), clopidogrel bisulfate (Plavix), etc.) 1 month prior to screening.
10. Acne scars that are considered post-inflammatory erythematous, post-inflammatory hyperpigmentation, varicella (chicken pox) scars, or perifollicular elastolysis will not be allowed to be identified as the target acne scars. These types of scars are still allowed to be present but cannot be selected.
11. Acne scars that are located in the glabella and temple regions. Acne scars located in these regions will not be allowed to be selected as a target or additional acne scar. As well, scars located in these areas will not be allowed to be treated during the study. Subjects are allowed to have acne scars located in these areas but cannot have them selected for evaluation or treated during the study.
12. Laser or light (red and blue) treatments for acne 3 months prior to screening.
13. Resurfacing procedures (CO2 , Erbium, Fraxel, etc.) performed 6 months prior to screening.
14. Any chemical peels in the last 30 days prior to screening.
15. Hypersensitivity to amid-type local anesthetics.
16. Any cortisol steroid or ILK injection 30 days prior to screening
17. Subjects with a history of diabetes.
18. Any medical condition or diagnosis which in the investigator's opinion would disqualify them from the research study.
19. History of abuse with the use of alcohol or drugs.
20. Participation in a clinical trial or use of an investigational product in the past 30 days.
21. Subjects who are considered health risks for participation in the study or the investigator determines not to be suitable.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
1 grade improvement of ASRS from baseline | Baseline-6 Months post first injection.
  The primary endpoint is a one grade improvement of the acne scar from baseline as rated on the ASRS.

SECONDARY OUTCOMES:
Statistically significant improvement of the acne scar from baseline | Baseline-6 Months post first injection.
  A significant improvement of the acne scar from baseline as rated by the
Statistically significant improvement of the skin quality from baseline | Baseline-6 Months post first injection.
  A significant improvement of the skin quality of the treatment area as rated by the investigator using the skin quality assessment scale.

OTHER OUTCOMES:
Statistically significant acne scar area reduction from baseline. | Baseline-6 Months post first injection.
  The first exploratory endpoint is a significant reduction of acne scar area as measured by the VECTRA system 6 months post first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Schweiger, M.D., Principal Investigator — CEO & Chief Medical Officer; Margaret J Tropeano, BS, Study Director — Clinical Research Director
Locations (1):
- Schweiger Dermatology, PLLC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is an investigator initiated study and will use the primary data to create a final data report. Individual patient data will not be available to other researchers.

REFERENCES:
- [Background] Fife D. Practical evaluation and management of atrophic acne scars: tips for the general dermatologist. J Clin Aesthet Dermatol. 2011 Aug;4(8):50-7. PMID 21909457
- [Background] Brandt FS, Cazzaniga A. Hyaluronic acid gel fillers in the management of facial aging. Clin Interv Aging. 2008;3(1):153-9. doi: 10.2147/cia.s2135. PMID 18488885
- [Background] Layton AM, Henderson CA, Cunliffe WJ. A clinical evaluation of acne scarring and its incidence. Clin Exp Dermatol. 1994 Jul;19(4):303-8. doi: 10.1111/j.1365-2230.1994.tb01200.x. PMID 7955470
- [Background] Koo JY, Smith LL. Psychologic aspects of acne. Pediatr Dermatol. 1991 Sep;8(3):185-8. doi: 10.1111/j.1525-1470.1991.tb00856.x. PMID 1836060
- [Background] Rivera AE. Acne scarring: a review and current treatment modalities. J Am Acad Dermatol. 2008 Oct;59(4):659-76. doi: 10.1016/j.jaad.2008.05.029. Epub 2008 Jul 26. PMID 18662839
- [Background] Tsao SS, Dover JS, Arndt KA, Kaminer MS. Scar management: keloid, hypertrophic, atrophic, and acne scars. Semin Cutan Med Surg. 2002 Mar;21(1):46-75. doi: 10.1016/s1085-5629(02)80719-2. No abstract available. PMID 11911537
- [Background] Jacob CI, Dover JS, Kaminer MS. Acne scarring: a classification system and review of treatment options. J Am Acad Dermatol. 2001 Jul;45(1):109-17. doi: 10.1067/mjd.2001.113451. PMID 11423843
- [Background] Sadick NS, Palmisano L. Case study involving use of injectable poly-L-lactic acid (PLLA) for acne scars. J Dermatolog Treat. 2009;20(5):302-7. doi: 10.1080/09546630902817879. PMID 19340629
- [Background] Lizzul PF, Narurkar VA. The role of calcium hydroxylapatite (Radiesse) in nonsurgical aesthetic rejuvenation. J Drugs Dermatol. 2010 May;9(5):446-50. PMID 20480786
- [Background] Brandt FS, Cazzaniga A. Hyaluronic acid fillers: Restylane and Perlane. Facial Plast Surg Clin North Am. 2007 Feb;15(1):63-76, vii. doi: 10.1016/j.fsc.2006.11.002. PMID 17317557
- [Background] Fife D, Zachary CB. Combining techniques for treating acne scars. Current Dermatology Reports. 2012;1:82-88.
- [Background] Werschler, Phillip, et al.
- [Background] Cohen JL. Understanding, avoiding, and managing dermal filler complications. Dermatol Surg. 2008 Jun;34 Suppl 1:S92-9. doi: 10.1111/j.1524-4725.2008.34249.x. PMID 18547189
- [Background] Hession MT, Graber EM. Atrophic acne scarring: a review of treatment options. J Clin Aesthet Dermatol. 2015 Jan;8(1):50-8. PMID 25610524
- [Background] Duranti F, Salti G, Bovani B, Calandra M, Rosati ML. Injectable hyaluronic acid gel for soft tissue augmentation. A clinical and histological study. Dermatol Surg. 1998 Dec;24(12):1317-25. doi: 10.1111/j.1524-4725.1998.tb00007.x. PMID 9865196
- [Background] Werschler, P. (2016). Severe - Depth = >2.5 mm in depth. Visibility = Substantial shadowing with tangential lighting. Journal of Drugs in Dermatology, 15(5), 518-525